CLINICAL TRIAL: NCT00422461
Title: A PHASE 2, RANDOMIZED, PLACEBO-CONTROLLED, DOSE-RANGING STUDY OF PF-00489791 IN SUBJECTS WITH STAGE 1 AND 2 ESSENTIAL HYPERTENSION USING AMBULATORY BLOOD PRESSURE MONITORING (ABPM)
Brief Title: A Dose Finding Study Of PF-00489791 In Patients With Mild To Moderate High Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A7331007
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Hypertension
Keywords: Clinical Trial; Randomized Controlled Trial; Humans; Cyclic Nucleotide Phosphodiesterases Type 5
MeSH Terms: conditions — Hypertension | interventions — PF-00489791

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- PF-00489791 20 mg titrated to 40 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 4 mg (Experimental)
  Interventions: Drug: PF-00489791
- PF-00489791 10 mg (Experimental)
  Interventions: Drug: PF-00489791

INTERVENTIONS:
Drug: placebo — placebo, oral, tablets, once daily, for 28 days
  Arms: Placebo
Drug: PF-00489791 — PF-00489791 20 mg titrated to 40 mg, oral, tablets, once daily, for 28 days
  Arms: PF-00489791 20 mg titrated to 40 mg
Drug: PF-00489791 — PF-00489791 4 mg, oral, tablets, once daily, for 28 days
  Arms: PF-00489791 4 mg
Drug: PF-00489791 — PF-00489791 10 mg, oral, tablets, once daily, for 28 days
  Arms: PF-00489791 10 mg

SUMMARY:
The purpose of this study is to evaluate the safety and blood pressure lowering effect of different doses of PF-00489791 in patients with mild to moderate high blood pressure

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or Females of non-childbearing potential between 18 and 70 years of age
2. History of mild to moderate hypertension

Exclusion Criteria:

1. Type 1 or 2 diabetes on prescribed medications
2. Secondary, severe, or malignant hypertension
3. History of a significant cardiovascular event within the last 12 months of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-02-27 (Actual); Primary Completion 2008-01-28 (Actual); Study Completion 2008-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- United States (20):
  - National Research Institute, Los Angeles, California
  - Apex Research Institute, Santa Ana, California
  - Orange County Research Center, Tustin, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Andres Patron, DO, PA, Pembroke Pines, Florida
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Twin Cities Clinical Research, Brooklyn Center, Minnesota
  - Riser Medical Associates, Picayune, Mississippi
  - Midwest Internists Clinical Research, P.C., St Louis, Missouri
  - Triangle Medical Research Associates, LLC, Cary, North Carolina
  - Medical Research Associates of Charlotte, Inc, Charlotte, North Carolina
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - Triangle Medical Research, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Sterling Research Group limited, Cincinnati, Ohio
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Clinical Research Associates Incorporated, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7331007&StudyName=A%20Dose%20Finding%20Study%20Of%20PF-00489791%20In%20Patients%20With%20Mild%20To%20Moderate%20High%20Blood%20Pressure

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 426 participants were screened, of whom 291 participants were screen failed and 135 participants were enrolled in the study and assigned to study treatment.
Groups:
- Placebo: Participants with mild to moderate hypertension were randomized to receive placebo orally, once daily for 28 days. Participants were followed up to maximum of 14 days after the last dose.
- PF-00489791 4 mg: Participants with mild to moderate hypertension were randomized to receive PF-00489791 4 milligram (mg) (2 tablets of 2 mg) orally, once daily for 28 days. Participants were followed up to maximum of 14 days after the last dose.
- PF-00489791 10 mg: Participants with mild to moderate hypertension were randomized to receive PF-00489791 10 mg tablet orally, once daily for 28 days. Participants were followed up to maximum of 14 days after the last dose.
- PF-00489791 20/40 mg: Participants with mild to moderate hypertension were randomized to receive PF-00489791 20 mg (2 tablets of 10 mg) orally, once daily for 14 days and then 40 mg (4 tablets of 10 mg) orally once daily for next 14 days. Participants were followed up to maximum of 14 days after the last dose.
Period: Overall Study
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Started | 35 | 35 | 32 | 33
Treated | 34 | 34 | 32 | 33
Full Analysis Set | 34 | 34 | 31 | 33
Completed | 32 | 32 | 31 | 30
Not Completed | 3 | 3 | 1 | 3
Not completed — Adverse Event | 1 | 2 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 2
Not completed — Participants no longer willing to participate in study | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who took at least 1 dose of study drug.
Groups:
- PF-00489791 4 mg: Participants with mild to moderate hypertension were randomized to receive PF-00489791 4 mg (2 tablets of 2 mg) orally, once daily for 28 days. Participants were followed up to maximum of 14 days after the last dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg | Total
Number analyzed (Participants) | 34 | 34 | 32 | 33 | 133
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 2 | 1 | 2 | 6 | 11
  45-64 years | 28 | 27 | 26 | 23 | 104
  Greater than or equal to (>=) 65 years | 4 | 6 | 4 | 4 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 13 | 10 | 49
  Male | 20 | 22 | 19 | 23 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Daytime Systolic Blood Pressure (SBP) as Measured by Ambulatory Blood Pressure Monitoring (ABPM) at Day 28
Description: The ABPM device was automatically programmed to inflate at every 20 minutes from 05:00 until 21:59 hours and from 22:00 to 04:59 hours the device inflated every 60 minutes. 24-hour clock time was used. ABPM was performed in this study on Baseline, Day 1, 14 and 28. Mean daytime SBP was an average of SBP measurements taken between 08:00 and 16:00 hours by ABPM device on the specified time points. In this outcome measure change from baseline in mean daytime SBP at Day 28 is reported.
Time Frame: From 08:00 to 16:00 hours on Baseline (Day 0, 1 day prior to first double-blind dose of study drug) and Day 28
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication and had a valid baseline and at least 1 valid post-baseline assessment of the primary endpoint. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 31 | 30 | 30 | 30
millimeter of mercury | 1.38 (1.55) | -1.42 (1.12) | -3.28 (1.08) | -5.59 (1.54)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 4 mg; Test type: Superiority; p = 0.0822, Nonlinear dose response regression model; Least square (LS) mean difference = -2.80, 95% CI 2-sided [-5.97 to 0.36], Standard Error of Mean 1.60
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 10 mg; Test type: Superiority; p = 0.0170, Nonlinear dose response regression model; LS mean difference = -4.66, 95% CI 2-sided [-8.47 to -0.85], Standard Error of Mean 1.92
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20/40 mg; Test type: Superiority; p = 0.0026, Nonlinear dose response regression model; LS mean difference = -6.97, 95% CI 2-sided [-11.45 to -2.48], Standard Error of Mean 2.26

2. Secondary Outcome: Change From Baseline in Mean Daytime Diastolic Blood Pressure (DBP) as Measured by ABPM at Day 28
Description: The ABPM device was automatically programmed to inflate at every 20 minutes from 05:00 until 21:59 hours and from 22:00 to 04:59 hours the device inflated every 60 minutes. 24-hour clock time was used. ABPM was performed in this study on Baseline, Day 1, 14 and 28. Mean daytime DBP was an average of DBP measurements taken between 08:00 and 16:00 hours by ABPM device on the specified time points. In this outcome measure change from baseline in mean daytime DBP at Day 28 is reported.
Time Frame: From 08:00 to 16:00 hours on Baseline (Day 0, 1 day prior to first double-blind dose of study drug) and Day 28
Population: FAS included all randomized participants who received at least 1 dose of study medication and had a valid baseline and at least 1 valid post-baseline assessment of the primary endpoint. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 31 | 30 | 30 | 30
millimeter of mercury | 0.73 (1.09) | -1.97 (0.81) | -3.83 (0.78) | -6.23 (1.09)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 4 mg; Test type: Superiority; p = 0.0264, Nonlinear dose response regression model; LS mean difference = -2.70, 95% CI 2-sided [-5.09 to -0.32], Standard Error of Mean 1.20
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 10 mg; Test type: Superiority; p = 0.0016, Nonlinear dose response regression model; LS mean difference = -4.56, 95% CI 2-sided [-7.35 to -1.77], Standard Error of Mean 1.41
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20/40 mg; Test type: Superiority; p < 0.0001, Nonlinear dose response regression model; LS mean difference = -6.96, 95% CI 2-sided [-10.03 to -3.89], Standard Error of Mean 1.55

3. Secondary Outcome: Change From Baseline in Mean 24-Hour SBP and DBP as Measured by ABPM at Day 28
Description: The ABPM device was automatically programmed to inflate at every 20 minutes from 05:00 until 21:59 hours and from 22:00 to 04:59 hours the device inflated every 60 minutes. 24-hour clock time was used. ABPM was performed in this study on Baseline, Day 1, 14 and 28. Mean 24-hour SBP and DBP was an average of SBP and DBP measurements, respectively, taken for 24 hours by ABPM device respectively. In this outcome measure change from baseline in mean 24-hour SBP and DBP at Day 28 is reported.
Time Frame: Over 24 hours on Baseline (Day 0, 1 day prior to first double-blind dose of study drug) and Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 30 | 30 | 28 | 29
millimeter of mercury
  SBP | -0.53 (1.53) | -0.40 (1.47) | -5.28 (1.55) | -3.96 (1.57)
  DBP | -0.13 (1.07) | -1.58 (1.07) | -3.94 (1.09) | -4.09 (1.09)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 4 mg; For SBP; Test type: Superiority; p = 0.9479, ANCOVA; LS mean difference = 0.13, 95% CI 2-sided [-3.79 to 4.05], Standard Error of Mean 1.98
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 10 mg; For SBP; Test type: Superiority; p = 0.0215, ANCOVA; LS mean difference = -4.75, 95% CI 2-sided [-8.78 to -0.72], Standard Error of Mean 2.03
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20/40 mg; For SBP; Test type: Superiority; p = 0.0886, ANCOVA; LS mean difference = -3.43, 95% CI 2-sided [-7.39 to 0.53], Standard Error of Mean 2.00
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 4 mg; For DBP; Test type: Superiority; p = 0.3173, ANCOVA; LS mean difference = -1.45, 95% CI 2-sided [-4.30 to 1.41], Standard Error of Mean 1.44
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 10 mg; For DBP; Test type: Superiority; p = 0.0087, ANCOVA; LS mean difference = -3.81, 95% CI 2-sided [-6.64 to -0.99], Standard Error of Mean 1.42
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 20/40 mg; For DBP; Test type: Superiority; p = 0.0062, ANCOVA; LS mean difference = -3.95, 95% CI 2-sided [-6.76 to -1.15], Standard Error of Mean 1.41

4. Secondary Outcome: Minimum and Maximum SBP and DBP as Measured by ABPM Over 24 Hours on Baseline, Day 1, 14 and 28
Description: The ABPM device was automatically programmed to inflate at every 20 minutes from 05:00 until 21:59 hours and from 22:00 to 04:59 hours the device inflated every 60 minutes. 24-hour clock time was used. ABPM was performed on Baseline, Day 1, 14 and 28. In this outcome measure maximum and minimum SBP and DBP values recorded by ABPM device over 24 hours on Baseline, Day 1, 14 and 28 are reported.
Time Frame: Over 24 hours on Baseline (Day 0, 1 day prior to first double-blind dose of study drug), Day 1, 14 and 28
Population: FAS included all randomized participants who received at least 1 dose of study medication and had a valid baseline and at least 1 valid post-baseline assessment of the primary endpoint. Here, "number analyzed" signifies participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 31 | 33
millimeter of mercury
  Maximum SBP: Baseline | 176.65 (12.38) | 179.68 (12.40) | 184.58 (15.30) | 177.45 (15.42)
  Maximum SBP: Day 1: number analyzed (Participants) | 32 | 33 | 29 | 32
  Maximum SBP: Day 1 | 173.13 (12.21) | 176.67 (19.60) | 175.62 (12.29) | 168.00 (12.17)
  Maximum SBP: Day 14: number analyzed (Participants) | 33 | 29 | 30 | 31
  Maximum SBP: Day 14 | 177.58 (14.53) | 177.90 (21.59) | 179.60 (11.75) | 176.52 (16.68)
  Maximum SBP: Day 28: number analyzed (Participants) | 30 | 30 | 28 | 29
  Maximum SBP: Day 28 | 177.33 (14.54) | 180.40 (19.40) | 177.04 (14.29) | 174.69 (12.14)
  Minimum SBP: Baseline | 117.88 (11.79) | 114.38 (12.65) | 122.52 (11.66) | 115.30 (13.60)
  Minimum SBP: Day 1: number analyzed (Participants) | 32 | 33 | 29 | 32
  Minimum SBP: Day 1 | 119.06 (12.32) | 110.27 (14.38) | 110.21 (13.46) | 109.38 (13.30)
  Minimum SBP: Day 14: number analyzed (Participants) | 33 | 29 | 30 | 31
  Minimum SBP: Day 14 | 113.82 (12.76) | 114.31 (13.59) | 114.07 (11.99) | 111.94 (10.52)
  Minimum SBP: Day 28: number analyzed (Participants) | 30 | 30 | 28 | 29
  Minimum SBP: Day 28 | 117.57 (15.54) | 114.27 (13.66) | 116.64 (10.28) | 110.34 (8.32)
  Maximum DBP: Baseline | 116.21 (7.01) | 114.53 (10.53) | 116.81 (11.97) | 116.76 (9.86)
  Maximum DBP: Day 1: number analyzed (Participants) | 32 | 33 | 29 | 32
  Maximum DBP: Day 1 | 113.81 (8.13) | 110.58 (10.29) | 111.38 (9.63) | 109.41 (11.16)
  Maximum DBP: Day 14: number analyzed (Participants) | 33 | 29 | 30 | 31
  Maximum DBP: Day 14 | 115.03 (9.17) | 111.97 (10.61) | 111.97 (10.35) | 111.58 (10.09)
  Maximum DBP: Day 28: number analyzed (Participants) | 30 | 30 | 28 | 29
  Maximum DBP: Day 28 | 117.20 (11.86) | 113.10 (9.42) | 112.32 (11.76) | 111.97 (10.58)
  Minimum DBP: Baseline | 68.15 (9.08) | 63.50 (8.31) | 67.90 (9.01) | 65.18 (8.11)
  Minimum DBP: Day 1: number analyzed (Participants) | 32 | 33 | 29 | 32
  Minimum DBP: Day 1 | 67.69 (9.30) | 60.67 (8.86) | 59.34 (8.52) | 60.16 (8.60)
  Minimum DBP: Day 14: number analyzed (Participants) | 33 | 29 | 30 | 31
  Minimum DBP: Day 14 | 65.48 (9.15) | 62.07 (9.51) | 61.13 (9.75) | 62.45 (8.20)
  Minimum DBP: Day 28: number analyzed (Participants) | 30 | 30 | 28 | 29
  Minimum DBP: Day 28 | 65.93 (11.58) | 62.23 (7.78) | 64.11 (8.71) | 61.38 (8.42)

5. Secondary Outcome: Change From Baseline in Cuff SBP and DBP at Day 28
Description: At Baseline and Day 28 visit, sitting cuff SBP and DBP was measured with the participant's arm supported at the level of the heart. The participant sat with feet flat on the floor for 5 minutes before the first BP was obtained. The BP measurement was done in duplicate approximately 5 minutes apart. The mean of duplicate measurements was recorded.
Time Frame: Baseline (pre dose value on Day 1 of treatment), Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 32 | 31 | 31 | 30
millimeter of mercury
  Cuff SBP | -4.60 (1.88) | -5.20 (1.82) | -4.97 (1.89) | -9.76 (1.95)
  Cuff DBP | -1.33 (1.27) | -4.37 (1.22) | -5.82 (1.27) | -5.63 (1.30)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 4 mg; For cuff SBP; Test type: Superiority; p = 0.8091, ANCOVA; LS mean difference = -0.60, 95% CI 2-sided [-5.51 to 4.31], Standard Error of Mean 2.48
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 10 mg; For cuff SBP; Test type: Superiority; p = 0.8809, ANCOVA; LS mean difference = -0.37, 95% CI 2-sided [-5.21 to 4.48], Standard Error of Mean 2.44
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20/40 mg; For cuff SBP; Test type: Superiority; p = 0.0382, ANCOVA; LS mean difference = -5.16, 95% CI 2-sided [-10.04 to -0.29], Standard Error of Mean 2.46
Statistical Analysis 4: Comparison: Placebo vs PF-00489791 4 mg; For cuff DBP; Test type: Superiority; p = 0.0731, ANCOVA; LS mean difference = -3.03, 95% CI 2-sided [-6.35 to 0.29], Standard Error of Mean 1.67
Statistical Analysis 5: Comparison: Placebo vs PF-00489791 10 mg; For cuff DBP; Test type: Superiority; p = 0.0077, ANCOVA; LS mean difference = -4.49, 95% CI 2-sided [-7.77 to -1.22], Standard Error of Mean 1.65
Statistical Analysis 6: Comparison: Placebo vs PF-00489791 20/40 mg; For cuff DBP; Test type: Superiority; p = 0.0111, ANCOVA; LS mean difference = -4.29, 95% CI 2-sided [-7.58 to -1.00], Standard Error of Mean 1.66

6. Secondary Outcome: Change From Baseline in Cuff SBP and DBP at Day 31
Description: At Baseline and Day 31 visit, sitting cuff SBP and DBP was measured with the participant's arm supported at the level of the heart. The participant sat with feet flat on the floor for 5 minutes before the first BP was obtained. The BP measurement was done in duplicate approximately 5 minutes apart. The mean of duplicate measurements was recorded.
Time Frame: Baseline (pre dose value on Day 1 of treatment), Day 31
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 31 | 32
millimeter of mercury
  Cuff SBP | 0.4 (10.18) | -0.6 (11.39) | -0.3 (10.96) | 0.4 (13.07)
  Cuff DBP | -0.7 (6.76) | -0.2 (7.47) | -0.8 (7.58) | 0.3 (7.86)

7. Secondary Outcome: Change From Baseline in Cuff Mean Arterial Pressure (MAP) at Day 28
Description: At Baseline and Day 28, sitting cuff MAP was measured with the participant's arm supported at the level of the heart. The participant sat with feet flat on the floor for 5 minutes before the first MAP was obtained. The MAP measurement was done in duplicate approximately 5 minutes apart. The mean of duplicate measurements was recorded.
Time Frame: Baseline (pre dose value on Day 1 of treatment), Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeter of mercury
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 32 | 31 | 31 | 30
millimeter of mercury | -2.59 (1.29) | -4.54 (1.26) | -5.53 (1.31) | -7.06 (1.34)
Statistical Analysis 1: Comparison: Placebo vs PF-00489791 4 mg; Test type: Superiority; p = 0.2567, ANCOVA; LS mean difference = -1.94, 95% CI 2-sided [-5.32 to 1.44], Standard Error of Mean 1.70
Statistical Analysis 2: Comparison: Placebo vs PF-00489791 10 mg; Test type: Superiority; p = 0.0860, ANCOVA; LS mean difference = -2.94, 95% CI 2-sided [-6.29 to 0.42], Standard Error of Mean 1.69
Statistical Analysis 3: Comparison: Placebo vs PF-00489791 20/40 mg; Test type: Superiority; p = 0.0103, ANCOVA; LS mean difference = -4.46, 95% CI 2-sided [-7.85 to -1.08], Standard Error of Mean 1.71

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study drug and up to 14 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and all non-SAEs.
Time Frame: Day 1 up to 14 days after last dose of study drug (maximum up to 42 days)
Population: Safety analysis set included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 32 | 33
Participants
  TEAEs | 12 | 11 | 11 | 13
  SAEs | 1 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for laboratory abnormalities included: hemoglobin, hematocrit, red blood cell count, total neutrophils, total protein, albumin: <0.8* limit of normal (LLN). Platelets: less than (<)0.5* LLN, greater than (>)1.75* upper limit of normal (ULN); white blood cell, glucose: <0.6*LLN, >1.5*ULN, lymphocytes: <0.8*LLN; >1.2*ULN; basophils, monocytes, eosinophils, total protein, albumin, uric acid: >1.2*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase: >3.0*ULN; blood urea nitrogen, creatinine: >1.3*ULN; sodium: <0.95*LLN, >1.05*ULN; potassium, chloride, calcium: <0.9*LLN, >1.1*ULN; creatine kinase: > 2.0*ULN, > 3.0*ULN, >10.0*ULN; total bilirubin, direct bilirubin, indirect bilirubin:>1.5*ULN; urinalysis: urine pH: <4.5, >8, glucose, ketones, protein, blood/hemoglobin: >=1, RBC, WBC, epithelial cells: >=6, casts: >1, bacteria: >20.
Time Frame: Day 1 up to 14 days after last dose of study drug (maximum up to 42 days)
Population: Safety analysis set included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 32 | 33
Participants | 10 | 9 | 11 | 10

10. Secondary Outcome: Change From Baseline in Heart Rate at Baseline, Day 1, 7, 14, 21, 28 and 31
Description: Sitting heart rate was measured with the participant's arm supported at the level of the heart. The participant sat with feet flat on the floor for 5 minutes before the heart rate was measured. The heart rate was measured for a minimum of 30 seconds, and the average of two measurements was recorded. Heart rate was measured in beats per minute.
Time Frame: Baseline (pre dose value on Day 1 of treatment), Day 1, 7, 14, 21, 28, 31
Population: FAS included all randomized subjects who received at least 1 dose of study medication and had a valid baseline and at least 1 valid post-baseline assessment of the primary endpoint. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 31 | 33
Beats per minute
  Baseline | 71.5 (8.76) | 69.2 (8.43) | 67.9 (8.63) | 68.3 (7.90)
  Change at Day1: number analyzed (Participants) | 25 | 28 | 26 | 26
  Change at Day1 | 0.5 (6.04) | 1.8 (6.64) | 4.8 (7.42) | 5.7 (8.14)
  Change at Day 7: number analyzed (Participants) | 34 | 33 | 31 | 33
  Change at Day 7 | -0.3 (5.92) | 1.5 (7.44) | 3.2 (9.60) | 4.6 (8.47)
  Change at Day 14: number analyzed (Participants) | 33 | 32 | 30 | 31
  Change at Day 14 | -1.2 (5.35) | -0.1 (8.08) | 1.6 (8.23) | 4.0 (7.15)
  Change at Day 21: number analyzed (Participants) | 32 | 32 | 30 | 30
  Change at Day 21 | 0.5 (7.27) | 2.9 (9.18) | -0.3 (8.55) | 4.9 (8.70)
  Change at Day 28: number analyzed (Participants) | 32 | 31 | 31 | 30
  Change at Day 28 | -0.0 (7.77) | 0.5 (7.78) | 0.8 (9.31) | 3.4 (9.38)
  Change at Day 31: number analyzed (Participants) | 34 | 34 | 31 | 32
  Change at Day 31 | -1.4 (8.85) | -0.3 (8.17) | 0.7 (8.76) | 4.8 (8.26)

11. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Following ECG parameters were evaluated: QT interval, QTc interval, RR interval, PR interval, QRS complex and heart rate. Clinical significant ECG findings were determined by the investigator's discretion.
Time Frame: Day 1 up to 14 days after last dose of study drug (maximum up to 42 days)
Population: Safety analysis set included all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
Number analyzed (Participants) | 34 | 34 | 32 | 33
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 14 days after last dose of study drug (maximum up to 42 days)
Description: Same event may appear as both an adverse events (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis set included all participants who took at least 1 dose of study drug.
Arm/Group | Placebo | PF-00489791 4 mg | PF-00489791 10 mg | PF-00489791 20/40 mg
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/34 | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 12/34 | 11/34 | 11/32 | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | PF-00489791 4 mg (N=34) | PF-00489791 10 mg (N=32) | PF-00489791 20/40 mg (N=33)
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | PF-00489791 4 mg (N=34) | PF-00489791 10 mg (N=32) | PF-00489791 20/40 mg (N=33)
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 2
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 7 | 6
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 1 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 1 | 1 | 1
Spontaneous penile erection (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.